CLINICAL TRIAL: NCT05906758
Title: Randomized Controlled Trial of Ultra-Low Contrast Coronary Angiography During Acute Kidney Injury (AKI)
Brief Title: Ultra-Low Contrast Angiography in AKI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-874
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: Coronary angiography; Ultra low contrast
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cerebral Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention arm (Active Comparator): Immediate angiography will be performed within 24 hours of enrollment. Omnipaque contrast will be administered. Serum creatinine will be collected on enrollment, within 6 hours before coronary angiography, and at 24h, 48h and 1-week after the angiography, as expected in common practice. Pre- and post-hydration administration will be at the discretion of the treating physician. In case percutaneous coronary intervention is indicated it will be schedule for 7 days after angiography.
  Interventions: Procedure: Angiography
- Delayed intervention arm (Placebo Comparator): Delayed angiography will be performed after kidney function stabilizes.
  Interventions: Procedure: Angiography

INTERVENTIONS:
Procedure: Angiography — Coronary angiography with less than 20cc of contrast materials

SUMMARY:
The aim of this study is to evaluate the safety of ultra-low contrast coronary angiography in patients with pre-existing acute kidney injury.

DETAILED DESCRIPTION:
The study is a non-inferiority open-label randomized controlled trial. Hospitalized patients who have AKI at admission or who develop AKI during admission and require invasive coronary angiography will be included in the trial. Once indication for invasive coronary angiography is determined, patients will be randomized to immediate angiography or to delayed angiography after renal function stabilizes. Immediate angiography will be performed within 24 of enrollment. Serum creatinine will be collected on enrollment, within 6 hours before coronary angiography, and at 24h, 48h and 1-week after the angiography, as expected in common practice. Pre- and post-hydration administration will be at the discretion of the treating physician. In case percutaneous coronary intervention is indicated it will be schedule for 7 days after angiography.

Definitions: AKI is defined as an increase in serum creatinine by ≥50% from baseline within 7 days or an increase in serum creatinine by ≥0.3 mg/dl within 2 days. CIN is defined as an increase in serum creatinine by 0.5mg/dl or a relative rise of 25% from the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who have AKI at admission or who develop AKI during admission and require invasive coronary angiography will be included in the trial.

Exclusion Criteria:

* Stabilized renal function manifested by unchanged or downtrending serum creatinine during a 24-hour period prior to enrollment.
* Contraindication for invasive coronary angiography other than AKI.
* Percutaneous coronary intervention is indicated and cannot be postponed by 7 days.
* Need for renal replacement therapy before coronary angiography or planned renal replacement therapy after coronary angiography (if premeditated before coronary angiography).
* Administration of intravascular contrast media during 7 days prior to the coronary angiography or within 6 days after coronary angiography.
* Pregnant patients, prisoners, cognitively impaired subjects, age below 18 years, unable or unwilling to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in incidence of Contrast Induced Nephropathy (CIN) | Within 7 days
  CIN is defined as an increase in serum creatinine by 0.5mg/dl or a relative rise of 25% from the baseline value. The investigators will measure the incidence of CIN by the increase in serum creatinine to see if the incidence will be the same in both arms whether the patient received the immediate angiography or if it was delayed until kidney function has been stabilized.

SECONDARY OUTCOMES:
Incidence of earlier occurrence of CIN | Within 7 days
  The investigators will measure serum creatinine at 24, 48 hours and at 1 week to measure if the occurrence of CIN will happen earlier in 1 arm than the other
Incidence of renal replacement therapy at up to 7 days post-angiography | Within 7 days
  The investigators will measure the incidence of renal replacement therapy by monitoring if the patient will undergo dialysis within 7 days post angiography

CONTACTS AND LOCATIONS:
Overall Officials: Zach Rozenbaum, MD, Principal Investigator — Tulane University
Locations (2):
- United States (2):
  - Tulane University Medical Center, New Orleans, Louisiana
  - University Medical Center, New Orleans, Louisiana